CLINICAL TRIAL: NCT06632587
Title: Comparing Outcomes Between Early and Standard-of-care Delayed Cranioplasty After Decompressive Hemicraniectomy
Brief Title: Timing Impact of Early vs. Late Cranioplasty on Hemicraniectomy Outcomes
Acronym: TIMELY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Pious Patel, Resident, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iRISID-2024-3103
Record Dates: First submitted 2024-09-26; First posted 2024-10-09 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-10

CONDITIONS: Craniocerebral Trauma; Stroke; Intracranial Hemorrhages
Keywords: Decompressive hemicraniectomy; cranioplasty; cranial trauma; stroke; intracranial hemorrhage; intracerebral hemorrhage; neurosurgery
MeSH Terms: conditions — Craniocerebral Trauma; Stroke; Intracranial Hemorrhages; Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The collection of outcomes will be performed without regard to the treatment versus control arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early cranioplasty (Active Comparator): Cranioplasty procedure performed prior to 8 weeks following the initial decompressive hemicraniectomy.
  Interventions: Procedure: Early cranioplasty
- Standard-of-care cranioplasty (Placebo Comparator): Cranioplasty procedure performed after 3 months following the initial decompressive hemicraniectomy.
  Interventions: Procedure: Standard-of-care cranioplasty

INTERVENTIONS:
Procedure: Early cranioplasty — Cranioplasty is the surgical procedure to restore the skull after a decompressive hemicraniectomy. The latter procedure is employed as a life-saving measure to relieve intracranial pressure in patients with acute cranial injuries. Early cranioplasty is defined as being performed within 8 weeks following the decompressive hemicraniectomy.
  Arms: Early cranioplasty
Procedure: Standard-of-care cranioplasty — Cranioplasty is the surgical procedure to restore the skull after a decompressive hemicraniectomy. The latter procedure is employed as a life-saving measure to relieve intracranial pressure in patients with acute cranial injuries. Standard-of-care cranioplasty is defined as being performed after 3 months following the decompressive hemicraniectomy.
  Arms: Standard-of-care cranioplasty

SUMMARY:
This prospective, randomized study aims to comprehensively evaluate the impact of cranioplasty timing on postoperative complications and long-term functional outcomes following decompressive hemicraniectomy (DHC). The primary endpoint focuses on comparing the rates of various postoperative complications, including infection, seizures, return to the operating room, and the need for ventriculoperitoneal shunting, between patients undergoing standard of care cranioplasty (>3 months after DHC) and those receiving early cranioplasty (within 8 weeks).

DETAILED DESCRIPTION:
This prospective, randomized study aims to comprehensively evaluate the impact of cranioplasty timing on postoperative complications and long-term functional outcomes following decompressive hemicraniectomy (DHC). The primary endpoint focuses on comparing the rates of various postoperative complications, including infection, seizures, return to the operating room, and the need for ventriculoperitoneal shunting, between patients undergoing standard of care cranioplasty (>3 months after DHC) and those receiving early cranioplasty (within 8 weeks).

The primary endpoint involves a comprehensive evaluation of long-term functional outcomes at 6 months post-injury ("injury" defined as "acute traumatic injury or source of increased intracranial pressure secondary to stroke or intracranial hemorrhage"). This assessment aims to determine whether the timing of cranioplasty influences patients' neurological recovery, cognitive function, and overall quality of life. By comparing the outcomes of patients who undergo standard of care cranioplasty with those who undergo early cranioplasty, the study seeks to provide valuable insights into the potential benefits of the latter approach.

The findings of this research hold the potential to guide clinical practice and inform decision-making for patients who have undergone DHC. By considering a range of complications and incorporating a robust statistical framework, the study contributes to a more nuanced understanding of the advantages and disadvantages associated with different cranioplasty timing strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adults of age greater than or equal to 18 years at the time of acute traumatic injury or source of increased intracranial pressure secondary to stroke or intracranial hemorrhage necessitating decompressive hemicraniectomy (DHC)
* Patient's cranial flap fulfills Craniectomy Contour Class A or B after 4 weeks postoperatively (doi:10.1227/ons.0000000000000689)
* Medically optimized for general anesthesia/surgery

Exclusion Criteria:

* Active systemic infection in weeks 6-8 post-DHC leading up to cranioplasty (e.g. pneumonia, urinary tract infection, soft tissue infection, bacteremia)
* Cranial infection in the post-DHC period
* Patient deemed not appropriate for early cranioplasty by attending neurosurgeon
* Patient mortality prior to 8 weeks post-injury ("injury" defined as "acute traumatic injury or source of increased intracranial pressure causing brain injury secondary to stroke or intracranial hemorrhage")

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcome at 6 months post-decompressive hemicraniectomy | 6 months post-decompressive hemicraniectomy
  modified Rankin scale outcome at 6 months post-decompressive hemicraniectomy
Functional outcome at 12 months post-decompressive hemicraniectomy | 12 months post-decompressive hemicraniectomy
  modified Rankin scale outcome at 12 months post-decompressive hemicraniectomy

SECONDARY OUTCOMES:
Post-cranioplasty seizure | 1 month post-cranioplasty
  Post-cranioplasty seizure occurrence, diagnosed clinically or on EEG
Post-cranioplasty hydrocephalus | 1 month post-cranioplasty
  Post-cranioplasty hydrocephalus or need for cerebrospinal fluid diversion
Post-cranioplasty return to operating room | 1 month post-cranioplasty
  All-cause return to operating room after cranioplasty
Post-cranioplasty infection | 12 months post-cranioplasty
  Surgical site or intracranial infection after cranioplasty
Post-cranioplasty disposition | 12 months post-cranioplasty
  Post-cranioplasty disposition (home, acute rehab, subacute rehab, death)
Post-cranioplasty length of hospital stay | 12 months post-cranioplasty
  Post-cranioplasty length of hospital stay
Readmission within 30 days post-cranioplasty | 30 days post-cranioplasty
  Readmission within 30 days post-cranioplasty

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospitals, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Patel PD, Khanna O, Gooch MR, Glener SR, Mouchtouris N, Momin AA, Sioutas G, Amllay A, Barsouk A, El Naamani K, Yudkoff C, Wyler DA, Jallo JI, Tjoumakaris S, Jabbour PM, Harrop JS. Clinical Outcomes After Ultra-Early Cranioplasty Using Craniectomy Contour Classification as a Patient Selection Criterion. Oper Neurosurg. 2023 Jul 1;25(1):72-80. doi: 10.1227/ons.0000000000000689. Epub 2023 May 5. PMID 37166197
- [Background] Malcolm JG, Rindler RS, Chu JK, Chokshi F, Grossberg JA, Pradilla G, Ahmad FU. Early Cranioplasty is Associated with Greater Neurological Improvement: A Systematic Review and Meta-Analysis. Neurosurgery. 2018 Mar 1;82(3):278-288. doi: 10.1093/neuros/nyx182. PMID 28419358
- [Background] Eaton JC, Greil ME, Nistal D, Caldwell DJ, Robinson E, Aljuboori Z, Temkin N, Bonow RH, Chesnut RM. Complications associated with early cranioplasty for patients with traumatic brain injury: a 25-year single-center analysis. J Neurosurg. 2022 Jan 21;137(3):776-781. doi: 10.3171/2021.11.JNS211557. Print 2022 Sep 1. PMID 35061995
- [Background] Sethi A, Chee K, Kaakani A, Beauchamp K, Kang J. Ultra-Early Cranioplasty versus Conventional Cranioplasty: A Retrospective Cohort Study at an Academic Level 1 Trauma Center. Neurotrauma Rep. 2022 Aug 1;3(1):286-291. doi: 10.1089/neur.2022.0026. eCollection 2022. PMID 36060455